CLINICAL TRIAL: NCT04435080
Title: Physical Rehabilitation in Intensive Care Unit in Acute Respiratory Distress Syndrome Patients With COVID-19
Brief Title: Physical Rehabilitation in ICU in ARDS Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.169.IRB1.037
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome; Rehabilitation; Intensive Care Unit Acquired Weakness; Critical Illness Polyneuromyopathy
Keywords: COVID-19; Acute Respiratory Distress Syndrome; Early rehabilitation; Intensive care unit acquired weakness
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-rehabilitation: The patients hospitalised in ICU who were provided all the intensive care managements except for rehabilitation interventions (discharged from intensive care unit before April 14, 2020)
- Rehabilitation: The patients hospitalised in ICU who were provided rehabilitation interventions in addition to all the intensive care managements. (discharged from intensive care unit after April 14, 2020)

SUMMARY:
The primary aim of this study is to evaluate the effect of physical rehabilitation performed in intensive care unit on the range of joint motions and muscle strength of survivors following discharge from intensive care unit in patients with COVID-19. Secondary outcome is to assess the duration of mechanical ventilation, length of stay in intensive care unit and in hospital, and mortality rates during intensive care unit stay and health related quality of life following discharge in survivors.

Until April 14 patients were provided all the intensive care managements except for rehabilitation and patients discharged before this time constituted the 'non-rehabilitation' group (n=17). Patients discharged after April 14 were provided rehabilitation in addition to usual intensive care unit care and constituted the study 'rehabilitation' group (n=18).

Passive range of motion exercises to each joint and neuromuscular electrical stimulation to bilateral quadriceps and tibialis anterior muscles were applied 6 days/week in the 'rehabilitation' group during intensive care unit stay.

DETAILED DESCRIPTION:
Patients with acute respiratory distress syndrome could develop muscle weakness associated with impairment of physical function defined as intensive care unit acquired weakness. Early rehabilitation is recommended to prevent complications including muscle weakness and joint contractures, enhance weaning from mechanical ventilation, improve outcome, quality of life.

COVID-19 is an acute infection with a high risk of enormous cytokine storm exacerbating the clinical condition in acute respiratory distress syndrome and is thought to further increase the risk of muscle weakness.

Study participants were recruited among patients hospitalized in the intensive care unit at Koc University Hospital. Standard care for these patients consisted of respiratory support, intravenous fluid therapy, medical treatment including anticoagulation and sedation, nutrition, change of position every 4 hours, and if needed, hemodynamic support. The non-rehabilitation group patients discharged before April 14, 2020, were provided with this standard care. The rehabilitation group patients that discharged after April 14, 2020, were provided rehabilitation in addition to usual standard care. The rehabilitation program consisted of a passive range of motion exercises for each joint of the extremities for 15 minutes/day, 6 days/week, and neuromuscular electrical stimulation to bilateral quadriceps and tibialis anterior muscles for 52 minutes/day, 6 days/week. The physiatrists evaluated the patients. Exercises and electrical stimulation were applied daily by physiotherapists. The physiatrist and anesthesiologist discussed the clinical status of the patients daily and the physiatrist modified the rehabilitation program, if needed. Patients were enrolled in the rehabilitation program if there is hemodynamical stability.

Information regarding demographic and clinical features, medications used, duration of mechanical ventilation, length of stay in the intensive care unit and hospital, and mortality were obtained from the digital patient records in both groups.

Following discharge, patients were evaluated for range of joint motion, manual muscle strength test, hand grip strength and Short form-36.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute respiratory distress syndrome secondary to COVID-19
* Hospitalised in intensive care unit
* Age older than 18 years

Exclusion Criteria:

* Acute respiratory distress syndrome due to other pathogens or causes
* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients that hospitalized due to acute respiratory distress syndrome secondary to COVID-19 were enrolled this study. The rehabilitation program was started at April 14, 2020 in intensive care unit. Until April 14, 2020 all patients were provided all the intensive care managements, except for rehabilitation. Therefore, patients discharged before this time constituted the 'non-rehabilitation' group of the present study. All patients discharged after April 14 were provided rehabilitation in addition to usual care and constituted the study 'rehabilitation' group
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 1 month after discharge from hospital
  Hand grip strength is an indicator of overall muscle strength that predicts mortality in older patients. Handgrip strength was measured using a handheld dynamometer according to the instructions of the American Society of Hand Therapists.Patients were seated placing their arms by their sides with the elbow flexed to 90°, the forearm mid-prone, and the wrist in neutral position. Patients were asked to grip the dynamometer with maximal effort using standard verbal encouragement. Three trials were performed in the dominant hand with a 30 sec rest between trials and the highest value was recorded in kg. The cut-off values of grip strength is 28.6 kg in men and 16.4 kg in women. The measurement was performed 1 month after discharge.

SECONDARY OUTCOMES:
Short form - 36 | 1 month after discharge from hospital
  Short form - 36 measures health related quality of life. It is a self-reported survey that evaluates individual health status with eight parameters consisting of physical function, pain, role limitations attributed to physical problems, role limitations attributed to emotional problems, mental health, social functioning, energy/ vitality, general health perception. There is not a summary score, each section is scored between 0-100, 0 indicates the worst condition, 100 indicates the best. The measurement was performed 1 month after discharge.
Length of stay in intensive care unit | through study completion, an average of 3 months
  Number of days of stay in intensive care unit from admission to discharge
Length of stay in hospital | through study completion, an average of 3 months
  Number of days of stay in hospital from admission to hospital to discharge from hospital
Duration of invasive mechanical ventilation | through study completion, an average of 3 months
  Number of days of invasive mechanical ventilation during intensive care unit
Manual muscle strength | 1 month after discharge from hospital
  Manual muscle strength was graded via a composite of Medical Research Council Scale score which has an excellent inter-rater reliability in survivors of critical illness. This scale range from 0 point (no muscle contraction) to 5 points (normal muscle strength). Through examination of 3 muscle groups in each limb (arm abduction, forearm flexion, wrist extension, hip flexion, knee extension and ankle dorsiflexion), clinical important muscle weakness has been defined as a composite score < 48 out of maximum 60 points. The measurement was performed 1 month after discharge.
Range of joint motion | 1 month after discharge from hospital
  Range of joint motion was evaluated in upper and lower extremity joints by physical examination and the results were recorded as normal or restricted for each joint. The measurement was performed 1 month after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozyemisci Taskiran, Prof, Principal Investigator — Koc University School of Medicine
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was not planned to share individual participant data

REFERENCES:
- [Result] Reid CL, Campbell IT, Little RA. Muscle wasting and energy balance in critical illness. Clin Nutr. 2004 Apr;23(2):273-80. doi: 10.1016/S0261-5614(03)00129-8. PMID 15030968
- [Result] Clavet H, Hebert PC, Fergusson D, Doucette S, Trudel G. Joint contracture following prolonged stay in the intensive care unit. CMAJ. 2008 Mar 11;178(6):691-7. doi: 10.1503/cmaj.071056. PMID 18332384
- [Result] Sosnowski K, Lin F, Mitchell ML, White H. Early rehabilitation in the intensive care unit: an integrative literature review. Aust Crit Care. 2015 Nov;28(4):216-25. doi: 10.1016/j.aucc.2015.05.002. Epub 2015 Jul 2. PMID 26142542
- [Result] Connolly B, O'Neill B, Salisbury L, Blackwood B; Enhanced Recovery After Critical Illness Programme Group. Physical rehabilitation interventions for adult patients during critical illness: an overview of systematic reviews. Thorax. 2016 Oct;71(10):881-90. doi: 10.1136/thoraxjnl-2015-208273. Epub 2016 May 24. PMID 27220357
- [Result] Walsh CJ, Batt J, Herridge MS, Dos Santos CC. Muscle wasting and early mobilization in acute respiratory distress syndrome. Clin Chest Med. 2014 Dec;35(4):811-26. doi: 10.1016/j.ccm.2014.08.016. Epub 2014 Sep 30. PMID 25453427
- [Result] Akar O, Gunay E, Sarinc Ulasli S, Ulasli AM, Kacar E, Sariaydin M, Solak O, Celik S, Unlu M. Efficacy of neuromuscular electrical stimulation in patients with COPD followed in intensive care unit. Clin Respir J. 2017 Nov;11(6):743-750. doi: 10.1111/crj.12411. Epub 2015 Dec 16. PMID 26597394
- [Result] Kleyweg RP, van der Meche FG, Schmitz PI. Interobserver agreement in the assessment of muscle strength and functional abilities in Guillain-Barre syndrome. Muscle Nerve. 1991 Nov;14(11):1103-9. doi: 10.1002/mus.880141111. PMID 1745285
- [Result] Turan Z, Ozyemisci Taskiran O, Erden Z, Kokturk N, Kaymak Karatas G. Does hand grip strength decrease in chronic obstructive pulmonary disease exacerbation? A cross-sectional study. Turk J Med Sci. 2019 Jun 18;49(3):802-808. doi: 10.3906/sag-1811-22. PMID 31190519
- [Result] Yoo JI, Choi H, Ha YC. Mean Hand Grip Strength and Cut-off Value for Sarcopenia in Korean Adults Using KNHANES VI. J Korean Med Sci. 2017 May;32(5):868-872. doi: 10.3346/jkms.2017.32.5.868. PMID 28378563
- [Result] Dodoo-Schittko F, Brandstetter S, Blecha S, Thomann-Hackner K, Brandl M, Knuttel H, Bein T, Apfelbacher C. Determinants of Quality of Life and Return to Work Following Acute Respiratory Distress Syndrome. Dtsch Arztebl Int. 2017 Feb 17;114(7):103-109. doi: 10.3238/arztebl.2017.0103. PMID 28302253